CLINICAL TRIAL: NCT04012671
Title: A Registered Cohort Study on Duchenne Muscular Dystrophy
Status: Recruiting | Type: Observational
Sponsor: Ning Wang, MD., PhD. (Other)
Responsible Party: Sponsor-Investigator, Ning Wang, MD., PhD., Professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAH of FMU [2019]193
Record Dates: First submitted 2019-07-07; First posted 2019-07-09 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-02

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dystrophinopathy is a term of X-linked recessive genetic disease, including Duchenne Muscular Dystrophy, Becker Muscular Dystrophy, and the X-linked dilated cardiomyopathy. The aim of this study is to determine the clinical spectrum and natural progression of dystrophinopathy in a prospective multicenter natural history study, to assess the clinical, genetic of patients with dystrophinopathy to optimize clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Beyond 2 years old
* Diagnosis with Duchenne Muscular Dystrophy, and female carriers, genotypically confirmed
* Diagnosis should be supported by muscle biopsy, if no genetic confirmation.

Exclusion Criteria:

* Presence of other clinically significant illness

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are diagnosed as Duchenne Muscular Dystrophy in the hosipital
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2039-12-31 (Estimated); Study Completion 2049-12-31 (Estimated)

PRIMARY OUTCOMES:
Age at death | 20 years
  the time when patient die

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, China